CLINICAL TRIAL: NCT04022486
Title: Seizures in Infants Hospitalized in Pediatric Intensive Care Unit for Bronchiolitis : Description and Risk Factors
Brief Title: Seizures in Infants Hospitalized in Pediatric Intensive Care Unit for Bronchiolitis
Acronym: BRONCHIOLITIS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: Bronchiolitis
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Bronchiolitis; Seizures; Hyponatremia
Keywords: Infant
MeSH Terms: conditions — Bronchiolitis; Seizures; Hyponatremia | interventions — Incidence; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children admitted in the PICU for severe bronchiolitis: Children admitted in the Pediatric Intensive Care Unit (PICU) for severe bronchiolitis between January 1st, 2010 and April 30th, 2018
  Interventions: Other: Incidence, management and risk factors of seizure

INTERVENTIONS:
Other: Incidence, management and risk factors of seizure — Incidence of seizure, management (treatment, paraclinical examinations) and risk factors of seizure in children admitted for severe bronchiolitis

SUMMARY:
Bronchiolitis is the leading cause of pediatric intensive care unit admission in infants. Seizures during bronchiolitis may be a neurological complication of respiratory viruses but also of the treatments. The investigating team's hypothesis is that the incidence of seizures is not so so uncommon in infants hospitalized in the pediatric intensive care unit for severe bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* age < 90 days
* hospitalization from January 1st, 2010 to April 30th, 2018 in the Pediatric Intensive Care Unit (PICU) of pediatric hospital in Lyon
* with bronchiolitis (clinical diagnosis according to American Academy of Pediatrics)

Exclusion Criteria:

* neurological history that may explain the occurrence of seizures
* significant congenital heart disease

Max Age: 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children hospitalized in the pediatric intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 805 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
: Incidence of seizure during bronchiolitis (before or during hospitalization in the pediatric intensive care unit) | Day 1
  Clinical or infra-clinical (diagnosed on Electroencephalography, EEG) seizure, simple or status epilepticus

CONTACTS AND LOCATIONS:
Overall Officials: Florent BAUDIN, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France